CLINICAL TRIAL: NCT05820087
Title: The HistoSonics Edison System for Treatment of Primary Solid Renal Tumors Using Histotripsy (#HOPE4KIDNEY US)
Brief Title: The HistoSonics Edison™ System for Treatment of Primary Solid Renal Tumors Using Histotripsy (#HOPE4KIDNEY)
Acronym: #HOPE4KIDNEY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP2083
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Renal Cancer; Tumor, Solid; Kidney Cancer; Tumor; Tumor, Benign
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, multi-center, single-arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HistoSonics Edison System (Experimental)
  Interventions: Device: HistoSonics Edison System

INTERVENTIONS:
Device: HistoSonics Edison System — Non-invasive destruction of kidney tissue using histotripsy, a non-thermal mechanical process of focused ultrasound.
  Other Names: Histotripsy

SUMMARY:
The purpose of this trial is to evaluate the effectiveness and safety of the HistoSonics Edison System for the destruction of kidney tissue by treating primary solid renal tumors.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, single-arm pivotal trial designed to evaluate the effectiveness and safety of the HistoSonics Edison System for the destruction of kidney tissue by treating primary solid renal tumors. Data through 90 days for all enrolled subjects will be summarized in a primary analysis to be submitted for Regulatory Submission to the FDA. Additionally, subjects will be followed for five (5) years post-index procedure, with evaluations at the 14-day, 30-day, 90-day, 180-day and annual time points.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥22 years of age.
2. Subject has signed the Institutional Review Board (IRB) approved trial Informed Consent Form (ICF) prior to any trial related tests/procedures and is willing to comply with trial procedures and required follow-up assessments.
3. Subject is diagnosed with only one (1) non-metastatic solid renal mass ≤3cm confirmed via CT or MRI ≤30 days prior to the index procedure date.
4. Subject has had a biopsy to determine the type of tumor, ≥14 days prior to the index procedure.
5. Subject can tolerate general anesthesia.
6. Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) grade 0-2 at baseline screening.
7. Subject meets all the following functional criteria at ≤14 days prior to the planned index procedure date:

   * White Blood Count (WBC) ≥3,000/mm3 (≥3 10*9/L)
   * Absolute Neutrophil Count (ANC) ≥1,200/mm3 (≥1.2 10*9/L)
   * Hemoglobin (Hgb) ≥9 g/dL
   * Platelet count ≥100,000/mm3 (≥100 10*9/L)
8. Subject has an eGFR (Glomerular filtration rate) ≥45mL/min, ≤14 days prior to the planned index procedure date.
9. The tumor selected for histotripsy treatment must be ≤3cm in longest diameter.
10. Subject has an adequate acoustic window to visualize targeted tumor using the HistoSonics Edison System.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant or nursing (lactating) during the trial period.
2. Subject is being actively treated in another pharmaceutical or device trial ≤30 days prior to planned index procedure date that may interfere with the primary endpoint(s).
3. Subjects who have active cancers (not in remission for the last two years) other than non-melanomatous skin cancers.
4. In the Investigator's opinion, the subject has co-morbid disease(s) or condition(s) that would cause undue risk and preclude safe use of the HistoSonics Edison System.
5. Subject is on dialysis, being considered for dialysis or has acute renal failure.
6. Subject has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or better from any adverse effects (except alopecia and neuropathy) related to previous therapy.
7. Subject has an International normalized ratio (INR) >1.5 or uncorrectable coagulopathy, (e.g., known von Willebrand disease, hemophilia, or on anticoagulants), on the planned index procedure date.
8. Subject is taking Aspirin (ASA) or NSAIDS ≤7 days prior to the planned index procedure date.
9. Subject has a life expectancy less than one (< 1) year.
10. In the investigator's opinion, histotripsy is not a treatment option for the subject.
11. Subject has a concurrent condition that could jeopardize the safety of the subject or compliance with the protocol.
12. Subject's targeted tumor has had prior locoregional therapy (e.g., ablation, embolization, radiation).
13. Subject's targeted tumor is not treatable by the HistoSonics Edison System's working ranges (refer to User Guide).
14. In the investigator's opinion, the anticipated risks of intervention outweigh the potential benefits of the intervention.
15. Subject has bilateral kidney tumors or has a single functioning kidney.
16. Subject has a genetic predisposition to kidney cancer such as:

    * Von Hippel Lindau (VHL)
    * Hereditary Papillary Renal Carcinoma (HPRC)
    * Birt-Hogg-Dubé Syndrome (BHD)
    * Tuberous Sclerosis Complex (TSC)
    * Hereditary Leiomyomata's Renal Cell Carcinoma (HLRCC)
    * Reed's Syndrome
    * Succinate Dehydrogenase B Deficiency (SDHB)
    * BRCA 1 associated protein -1 (BAP1) Renal Cell Carcinoma
    * MITF predisposed Renal Cell Carcinoma
17. The targeted tumor is an angiomyolipoma.
18. Subject has a known sensitivity to contrast media and cannot be adequately pre-medicated.
19. Subject has a urinary tract infection (UTI) ≤7 days prior to the planned index procedure date.
20. The targeted tumor is not clearly visible with ultrasound, MRI or CT.
21. Targeted tumor with adequate margin overlaps the renal pelvis, main renal vessel, ureter, organ or other vital structure.
22. The treatment of the tumor will not allow an adequate margin (as determined by the investigator).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Primary technique efficacy defined as the percentage of targeted tumors that were successfully eliminated after a single histotripsy session as assessed by contrast enhanced MRI or CT at 90 days. | 90 days Post Index Procedure
  Primary Effectiveness Endpoint
Primary Safety Endpoint - Freedom from index procedure related major complications, defined by Clavien-Dindo Classification Grade 3 or higher up to 30 days after the histotripsy procedure. | 30 days Post Index Procedure
  Primary Safety Endpoint

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint- Technical success demonstrating complete coverage of the targeted tumor as determined post-index procedure (≤36 hours) by contrast enhanced MRI or CT in subjects whom treatment was initiated. | Up to 36 hours Post Index Procedure
  Secondary Effectiveness Endpoint - Technical success defined as completion of histotripsy treatment according to protocol and demonstrating complete coverage of the targeted tumor as determined post-index procedure (≤36 hours) by contrast enhanced MRI or CT in subjects whom treatment was initiated.
Secondary Safety Endpoint - Freedom from index procedure related major complications, defined by Clavien-Dindo Classification Grade 3 or higher up to 90 days after the histotripsy procedure. | 90 days Post Index Procedure
  Secondary Safety Endpoint

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Providence Mission Hosptial, Mission Viejo, California
  - Yale School of Medicine, New Haven, Connecticut
  - AdventHealth Celebration, Celebration, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Northwell Health, Lake Success, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No